CLINICAL TRIAL: NCT00928356
Title: A Single Center Clinical Evaluation of Same Sitting Hybrid Revascularization: Robotic Coronary Artery Bypass Grafting and Percutaneous Coronary Intervention for the Treatment of Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pinnacle Health Cardiovascular Institute (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Same Sitting Robotic CABG/PCI
Record Dates: First submitted 2009-06-23; First posted 2009-06-25 (Estimated); Last update posted 2020-05-11 (Actual); Status verified 2019-03

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Robotic Coronary Artery Bypass Surgery; Percutaneous Coronary Intervention; Hybrid Coronary Revascularization
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hybrid CABG/PCI (Experimental): Patients undergo hybrid, same sitting CABG/PCI as described.
  Interventions: Procedure: Hybrid CABG/PCI
- Off-pump CABG (Other): Standard of Care Off Pump CABG
  Interventions: Procedure: Off Pump CABG

INTERVENTIONS:
Procedure: Hybrid CABG/PCI — Same sitting hybrid, robotic CABG/PCI
  Arms: Hybrid CABG/PCI
Procedure: Off Pump CABG — Standard of Care Off Pump CABG
  Arms: Off-pump CABG

SUMMARY:
The primary objective of this study is to assess the safety and effectiveness of same sitting, simultaneous hybrid robotic assisted coronary artery bypass grafting (CABG) and percutaneous coronary intervention (PCI) in the treatment of obstructive multivessel coronary artery disease. A secondary objective is the assessment and standardization of optimal operator techniques and comparative study of patients undergoing CABG during study period.

DETAILED DESCRIPTION:
The study population will consist of patients with multivessel coronary artery disease requiring CABG with suitable anatomy for combination CABG and PCI of non-bypassed arteries.

The primary endpoint of this feasibility study is a 30-day composite of major adverse clinical events including death, repeat revascularization, stroke and/or myocardial infarction.

The secondary endpoints include:

1. Successful completion of same sitting CABG and coronary stent procedure
2. Successful completion of CABG and PCI during single hospitalization
3. Achievement of complete revascularization
4. Patency of the LIMA and stented vessels as determined by coronary angiography at time of procedures or prior to discharge and by cardiac Computed Tomographic Angiography (CTA) or coronary angiography at 1 year.
5. Stent thrombosis at 24 hours (acute), 30 days (sub acute), and 1 year (late)
6. One-year composite clinical event endpoints of major clinical events including death, repeat revascularization, myocardial infarction, and freedom from angina
7. Comparative analysis of hospital, 30 day, and 1 year events of hybrid CABG patients compared to consecutive patients undergoing off pump CABG with standard thoracotomy during study period

ELIGIBILITY:
Inclusion Criteria:

* Requirement for CABG
* Anatomy and body habitus suitable for Robotic CABG
* Requirement of revascularization of arteries amendable for PCI but not accessable by Robotic CABG

Exclusion Criteria:

* Need for emergent CABG

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2008-10-14 (Actual); Primary Completion 2015-05-19 (Actual); Study Completion 2019-08-13 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this feasibility study is a 30-day composite of major adverse clinical events including death, repeat revascularization, stroke and/or myocardial infarction. | 1 year

SECONDARY OUTCOMES:
One-year composite clinical event endpoints of major clinical events. Comparative analysis of consecutive patients undergoing off pump CABG with standard thoracotomy during study period. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: William Bachinsky, M.D., Principal Investigator — Pinnacle Health Cardiovascular Institute, Inc.
Locations (1):
- UPMC Pinnacle Harrisburg, Harrisburg, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No